CLINICAL TRIAL: NCT01312558
Title: The Effect of the Mediterranean Diet on Obstructive Sleep Apnoea-Hypopnoea Syndrome: A Randomised Trial
Acronym: MEDOSAHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Christopher Papandreou, Christopher Papandreou, University of Crete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT01312558
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Obstructive Sleep Apnoea; Hypopnoea Syndrome
Keywords: obstructive sleep apnoea/hypopnoea syndrome; Mediterranean diet; exercise; weight loss; continuous positive airway pressure; lipid peroxidation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prudent diet group (Experimental): Participants follow CPAP therapy, a prudent diet while receiving counselling to increase their physical activity.
  Interventions: Behavioral: Prudent diet group
- Mediterranean diet group (Experimental): Participants follow CPAP therapy, Mediterranean diet, while receiving counselling to increase their physical activity.
  Interventions: Behavioral: Mediterranean diet group

INTERVENTIONS:
Behavioral: Prudent diet group
  Arms: Prudent diet group
Behavioral: Mediterranean diet group
  Arms: Mediterranean diet group

SUMMARY:
This study aims to investigate the role of the Mediterranean diet in obese patients with Obstructive sleep apnoea-hypopnoea syndrome.

DETAILED DESCRIPTION:
Obstructive sleep apnoea-hypopnoea syndrome (OSAHS) is considered to be one of the most prevalent sleep-related breathing disorders, with an enormous effect on public health. Approximately 2-4% of the general adult population experiences some degree of this syndrome. This percentage increases even more with obesity, up to 20-40%, especially in individuals with an excessive body mass index (BMI) > 30 kg/m2. OSAHS is associated with significant systemic consequences, including cardiovascular morbidity and mortality, and the risk increases with the severity of the syndrome. The pathophysiology underlying the link between OSAHS and the cardiovascular system is attributed largely to systemic inflammation and oxidative stress, which are both contributors to endothelial dysfunction. The treatment modalities of OSAHS include continuous positive airway pressure (CPAP), weight loss, upper airway surgery, and medication. CPAP is the first line therapy, as a means of maintaining upper airway patency, and it is well known that this intervention reduces morbidity and mortality. In severe cases of OSAHS the weight loss strategy is essential and must accompany CPAP treatment. A growing body of evidence in OSAHS supports the beneficial role of weight reduction, induced by diet alone or in combination with exercise, leading to a reduction in apnoeas and hypopnoeas.We aim to evaluate the effect of the Mediterranean diet compared with that of a prudent diet on obese OSAHS patients who were treated with CPAP while receiving counselling to increase their physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with apnoea-hypopnoea index >15/h and Epworth Sleepiness Scale > 10

Exclusion Criteria:

* Diseases such as ischaemic heart disease, diabetes mellitus, thyroid disorders, and malignancies
* Upper airway surgery
* Gestation
* Alcoholism
* Diet for weight reduction during the last 6 months
* Eating habits close to the Mediterranean diet at the entry phase
* Intake of antioxidant supplements
* Medications affecting weight
* Smoking (in the case of TBARS)
* Therapy with sleeping pills
* Use of anti-depressive medication
* BMI < 30.0 Kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
OSAS severity
  The primary outcome measure was the change in OSAS severity as reflected mainly by AHI and saturation indexes.

SECONDARY OUTCOMES:
AHI during REM sleep and lipid peroxidation marker TBARS

OTHER OUTCOMES:
Anthropometric measurements
  weight, height, waist circumference and neck circumference

CONTACTS AND LOCATIONS:
Locations (1):
- University of Crete, Heraklion, Greece

REFERENCES:
- [Derived] Papandreou C, Hatzis CM, Fragkiadakis GA. Effects of different weight loss percentages on moderate to severe obstructive sleep apnoea syndrome. Chron Respir Dis. 2015 Aug;12(3):276-8. doi: 10.1177/1479972315587516. Epub 2015 May 25. No abstract available. PMID 26015461
- [Derived] Papandreou C, Schiza SE, Bouloukaki I, Hatzis CM, Kafatos AG, Siafakas NM, Tzanakis NE. Effect of Mediterranean diet versus prudent diet combined with physical activity on OSAS: a randomised trial. Eur Respir J. 2012 Jun;39(6):1398-404. doi: 10.1183/09031936.00103411. Epub 2011 Oct 27. PMID 22034645
- [Derived] Papandreou C, Schiza SE, Tzatzarakis MN, Kavalakis M, Hatzis CM, Tsatsakis AM, Kafatos AG, Siafakas NM, Tzanakis NE. Effect of Mediterranean diet on lipid peroxidation marker TBARS in obese patients with OSAHS under CPAP treatment: a randomised trial. Sleep Breath. 2012 Sep;16(3):873-9. doi: 10.1007/s11325-011-0589-7. Epub 2011 Sep 15. PMID 21918812